CLINICAL TRIAL: NCT01880619
Title: A Randomized Clinical Trial Comparing Alpha Blacker (Tamsulosin) and Anticholinergic (Solifenacin) in Treatment of Ureteral Stent Related Symptoms
Brief Title: Comparison of Tamsulosin and Solifenacin in Treatment of Ureteral Stent Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment of USS
Record Dates: First submitted 2013-06-13; First posted 2013-06-19 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-08

CONDITIONS: Relieve of Ureteral Stent Symptoms
Keywords: Double J; Ureteral stents; Symptoms; Alpha blockers; Anticholinergic
MeSH Terms: interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Placebo Comparator): Patients in this group will receive placebo
  Interventions: Drug: Control
- Group B (Active Comparator): Patients in this group will receive Tamsulosin
  Interventions: Drug: Tamsulosin
- Group C (Active Comparator): Patients in this group will receive Solifenacin
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Tamsulosin — Patients in this arm will receive Tamsulosin 0.4 mg daily
  Other Names: Tamsulin
  Arms: Group B
Drug: Solifenacin — Patients in the arm will receive Solifenacin
  Other Names: Sofinacin
  Arms: Group C
Drug: Control — Patients in this are will receive placebo
  Arms: Group A

SUMMARY:
This study will be conducted to compare the effectiveness of alpha blocker (Tamsulosin) and Anticholinergic (Solifenacin) in relieving lower urinary tract symptoms caused DJ ureteral stents.

DETAILED DESCRIPTION:
Eligible patients who signed the informed consent will randomly assigned to one of 3 groups; group 1 (control), group 2 (tamsulosin) and group 3 (Solifenacin). Ureteral stent symptom questionnaire (USSQ) will be used to compare health related quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

Patient who will undergo unilateral ureteral stent fixation:

1. To relieve upper urinary tract obstruction caused by ureteric calculi
2. After ureteroscopic lithotripsy for ureteral calculi.

Exclusion Criteria:

1. Patients who had LUTS before stent fixation.
2. Ureteral stent fixation after open or laparoscopic surgery.
3. Bilateral ureteral stents.
4. Patients who developed complications related to the primary endoscopic procedure
5. Patients who developed stent related complications such as hematuria, acute pyelonephritis or stent displacement

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The Efficacy of tamsulosin and solifenacin in relieving ureteral stent symptoms will be evaluated by comparing the scores of ureteral stent symptoms questionnaire in the studied groups | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R EL-Nahas, A. Professor, Principal Investigator — Urology and Nephrology Center, Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

REFERENCES:
- [Derived] El-Nahas AR, Tharwat M, Elsaadany M, Mosbah A, Gaballah MA. A randomized controlled trial comparing alpha blocker (tamsulosin) and anticholinergic (solifenacin) in treatment of ureteral stent-related symptoms. World J Urol. 2016 Jul;34(7):963-8. doi: 10.1007/s00345-015-1704-3. Epub 2015 Oct 9. PMID 26453222